CLINICAL TRIAL: NCT02692521
Title: Human Milk Feeding Rates Post-NICU Discharge
Status: Completed | Type: Observational
Sponsor: Pediatrix (Other)
Responsible Party: Sponsor
Other Study IDs: PDX-001-15
Record Dates: First submitted 2016-02-17; First posted 2016-02-26 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Human Milk/Breastfeeding
MeSH Terms: interventions — Milk, Human

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Dietary Supplement: Human Milk

SUMMARY:
The purpose of this study is to discover the incentives and barriers to human milk use and breast-feeding in the NICU graduate. By better understanding the incentives and barriers we believe we can define better methods for promoting higher rates and longer duration of human milk use in this medically fragile population.

DETAILED DESCRIPTION:
The AAP continues to reaffirm its recommendation of exclusive breast feeding for about 6 months, with continuation of breastfeeding as complementary feeding starts. Ideally, breastfeeding continues for the first year of life. NICUs have implemented increasing use of human milk with reports of more than 80 percent of infants receiving at least some human milk at discharge. Research has shown that breastfeeding rates in preterm infants and initiation of breastfeeding at discharge are far less than that of term infants (Mastrup, 2014). Yet studies continue to show the ongoing benefits of breast milk initiation in low birth weight neonates while they are in the NICU and better developmental outcomes at 30 months of age (Vohr, Poindexter, Dusick, McKinley, et al., 2007). A large cohort of low birth weight infants studied revealed that those who were given breast milk early in their hospitalization and continued receiving it , whether expressed or breast fed, had less frequent re-hospitalizations and higher Bayley Developmental scores for emotional regulation at 30 months of age. Additionally, as their breast milk volume exposure increased, these children had improved mental development index and total behavioral index improvement as well.

In a CQI survey done in three NICU follow up clinics, we discovered that only about 30 percent were still breastfeeding at 1-3 months post discharge. There are a few studies investigating factors which contribute to increased human milk post discharge. Factors studied include kangaroo care, quick access to pumping support, and history of breast feeding while in the NICU.

There are a few studies investigating factors which contribute to increased human milk use post discharge. Callen and Pinelli found that successful breast feeding in preterm infants (mean gestation 28 weeks) was more likely in mothers who pumped early and continued diligently. In addition to early pumping and lactation support, kangaroo care, and having the experience of breast feeding while still in the NICU have been associated with longer use of human milk and successful breast feeding after discharge. Pineda (2011) looked at the effects of breast-feeding while in the NICU and whether the first oral sucking feeding was at the breast in preterm infants. Mean gestational age when the infant was put to breast was 33.1 weeks + 1.59 weeks. Though challenging for mothers, the ability to continue to maintain breast-feeding during the NICU stay and until discharge as well as having the first feed be at the breast increased overall duration of breast-feeding duration after discharge. Direct breast-feeding also increases oxytocin levels in the mother, which leads to psychological benefits such as improved maternal response and improved attachment behaviors. These factors may indirectly lead to improved use of breast milk.

This study will investigate which babies are receiving human milk, either expressed or breast fed at varying times post discharge, and further explores NICU factors which may foster or inhibit increasing breast milk use in NICU graduates.

ELIGIBILITY:
Inclusion Criteria:

* Survival to discharge
* Site ability to plan and implement developmental follow-up for two years corrected age

Exclusion Criteria:

* Parents unwilling to participate in follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: NICU Graduates
Sampling Method: Non-Probability Sample
Enrollment: 1160 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-02-03 (Actual)

PRIMARY OUTCOMES:
Identify barriers and incentives to the use of human milk in infants hospitalized in a NICU | 2 years
  Increase human milk use in post-NICU neonates by identifying barriers and incentives to the use of human milk in infants hospitalized in a NICU in order to maximize its use.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Ellis, MD, Principal Investigator — Pediatrix
Locations (5):
- United States (5):
  - Developmental Follow-up Clinic - Scottsdale / Kidz Clinic II, Scottsdale, Arizona
  - Summerlin Developmental Clinic, Las Vegas, Nevada
  - Dallas Developmental Pediatrics, Dallas, Texas
  - San Antonio Pediatric Development Services, San Antonio, Texas
  - Preemie Place High Risk Infant Follow-up Clinic, The Woodlands, Texas

REFERENCES:
- [Background] Briere CE, McGrath J, Cong X, Cusson R. An integrative review of factors that influence breastfeeding duration for premature infants after NICU hospitalization. J Obstet Gynecol Neonatal Nurs. 2014 May-Jun;43(3):272-81. doi: 10.1111/1552-6909.12297. Epub 2014 Apr 1. PMID 24689979
- [Background] Davanzo R, Ronfani L, Brovedani P, Demarini S; Breastfeeding in Neonatal Intensive Care Unit Study Group. Breast feeding very-low-birthweight infants at discharge: a multicentre study using WHO definitions. Paediatr Perinat Epidemiol. 2009 Nov;23(6):591-6. doi: 10.1111/j.1365-3016.2009.01068.x. PMID 19840296
- [Background] Furman L, Minich N, Hack M. Correlates of lactation in mothers of very low birth weight infants. Pediatrics. 2002 Apr;109(4):e57. doi: 10.1542/peds.109.4.e57. PMID 11927730
- [Background] Paula P. Meier, RN, DNSc, FAAN, Janet L. Engstrom, RN, PhD, CNM, WHNP-BC, Aloka L. Patel, MD, Briana J. Jegier, PhD, and Nicholas E. Bruns, Improving the Use of Human Milk During and After the NICU Stay. BSPublished online February 27, 2012 4Pediatrics Vol. 129 No. 3 March 1, 2012 pp. e827-e841 doi: 10.1542/peds.2011-3552
- [Background] Section on Breastfeeding. Breastfeeding and the use of human milk. Pediatrics. 2012 Mar;129(3):e827-41. doi: 10.1542/peds.2011-3552. Epub 2012 Feb 27. PMID 22371471
- [Derived] Fenrich AL, Shmorhun DP, Martin GC, Young JA, Cohen MI, Kelleher AS, Anyebuno MA, Rider ED, Motta CL, Clark RH. Long QT and Hearing Loss in High-Risk Infants Prospective Study Registry. Pediatr Cardiol. 2022 Dec;43(8):1898-1902. doi: 10.1007/s00246-022-02939-4. Epub 2022 Jun 3. PMID 35661239